CLINICAL TRIAL: NCT04203407
Title: Effects of a Culturally-sensitive Theory-driven Advance Care Planning (ACP) Game on Self-efficacy and ACP Behaviors Among Chinese Older Adults: a Mixed Method Study
Brief Title: Effects of a Culturally-sensitive Theory-driven Advance Care Planning (ACP) Game Among Chinese Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Xihu community healthcare service centre (Unknown); Guanshaling community healthcare service centre (Unknown)
Responsible Party: Principal Investigator, LIU Li, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CREC2019428; ChiCTR1900028190 (Registry Identifier: Chinese Clinical Trial Registry, ChiCTR)
Record Dates: First submitted 2019-12-15; First posted 2019-12-18 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Advance Care Planning; Game; Older Adults

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACP game (Experimental): Participants in the intervention group will be divided into groups of 4 participants to play a 1-hour culturally-sensitive theory-driven ACP board game with 15-minute debriefing delivered by facilitators. The ACP board game is developed by the principle investigator in a previous project.
  Interventions: Behavioral: ACP game
- Usual care (Active Comparator): Participants in the control group will receive a 1-hour board game about health lifestyle.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: ACP game — Participants in the intervention group will be divided into groups of 4 participants to play a 1-hour culturally-sensitive theory-driven ACP board game with 15-minute debriefing delivered by facilitators. The ACP board game is developed by the principle investigator in a previous project.
  Arms: ACP game
Behavioral: Usual care — Participants in the control group will receive a 1-hour board game about health lifestyle.
  Arms: Usual care

SUMMARY:
This proposed study aims to examine the effects of a culturally-sensitive theory-driven advance care planning (ACP) game in increasing the self-efficacy and readiness of ACP behaviours among Chinese community-dwelling older adults. This is a mixed methods study with the quantitative paradigm being the main research approached used. The quantitative arm will be a randomized controlled trial (RCT). The qualitative arm will adopt focus group interviews for data collection. Recruited subjects from the community centres will be randomly allocated to the intervention and control group. The older adults in the experimental group will receive an ACP board game delivered by trained facilitators, whereas the older adults in the control group will receive another board game about healthy lifestyle. The outcome measures of the older adults will include the ACP Engagement scale, the Life-Support Preferences Questionnaire (LSPQ), a self-developed ACP knowledge questionnaire and those data will be collected at baseline (T0), immediately post-intervention(T1), at 1 month (T2), and 3 month (T3). The qualitative arm of this study will contribute to the understanding of issues and effects of ACP game as an intervention. Its finding will complement the results obtained from the RCT.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years or over;
* speak Chinese.

Exclusion Criteria:

* uncommunicable because of language barrier or sensory impairment;
* have been referred to the palliative care service at the time of recruitment.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-08-08 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Advance Care Planning Engagement Scale | 3 months
  Behaviour changes in ACP behaviours measured using Advance Care Planning Engagement Scale. It is about different ACP behavior on a 5-point Likert scale. The higher score means the higher level of self-efficacy and readiness for the behaviours.

SECONDARY OUTCOMES:
Certainty rate of end-of-life preferences toward medical care | 3 months
  End-of-life preferences is measured by the Life-Support Preferences Questionnaire (LSPQ). It describes one hypothetical terminally ill scenario. Preferences regarding (i) three kinds of life-sustaining treatments (cardiopulmonary resuscitation, mechanical ventilator and tube feeding) based on three options (want to attempt, refuse or uncertain) and (ii) care goals (comfort-oriented, prolongation of life at all costs or uncertain) , will be asked.
Self-develped ACP knowledge questionnaire | 3 months
  The questionnaire comprised 10 questions. Response options for each of these questions were "yes" and "no". Content validity was assessed within a palliative care expert team.

OTHER OUTCOMES:
Change of emotional status | Immediate post-intervention
  Emotional status is measured using the Chinese version of the 7-item Generalized Anxiety Disorder ( GAD-7) scale as process indicators. The total score ranges from 0 to 21. Higher scores indicate higher level of anxiety.
Experience of playing ACP game | Immediate post-intervention
  Participants' experience of playing ACP game will be collected by focus group interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Li LIU, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Xihu community, guanshaling community, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No